CLINICAL TRIAL: NCT03484884
Title: A Feasibility Study of Non-Invasive Cerenkov Luminescence Imaging in Patients With Cancer
Brief Title: A Study of Optical Imaging With Light From Radiotracers in Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17-538
Record Dates: First submitted 2018-03-20; First posted 2018-04-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Cancer
Keywords: nodal metastases; 17-538; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thyroid cancer/nodal metastasis: Participants will have thyroid cancer and nodal metastasis in the neck, supraclavicular, axillary and/or inguinal area.
  Interventions: Diagnostic Test: Cerenkov luminescence imaging.

INTERVENTIONS:
Diagnostic Test: Cerenkov luminescence imaging. — Cerenkov luminescence imaging will be obtained from MSKCC patients who are scheduled for routine FDG PET scan or 131I therapy that emit a continuum of ultraviolet and visible light from the decay of certain radionuclides.

SUMMARY:
The purpose of this study is to test Cerenkov luminescence imaging, which is a different way to take pictures of thyroid cancer and/or any tumors with (existing or suspected) nodal metastases in the neck, supraclavicular, axillary and/or inguinal region.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 years of age or old
* Participant must meet one of the following:

  * Patients with thyroid cancer scheduled for thyroid ablation therapy with 131I
  * Patients with any tumors with (existing or suspected) nodal metastases in the neck, supraclavicular, axillary and/or inguinal region who are scheduled to receive a clinical FDG PET/CT scan
  * Patients with metastatic prostate cancer who are schedule for Xofigo therapy with 223Ra
  * Patients scheduled to receive a standard of care 66Ga-DOTA-TATE or [18f]-PARPi PET scan in the Nuclear Medicine Clinic
  * Patient undergoing Lu-DOTA TATE treatment in the Nuclear Medicine Clinic

Exclusion Criteria:

* Patients imaged for Cerenkov luminescence are going to be required to be in a darkened enclosure for at least 10 minutes and sit still during image acquisition. Any conditions that would prevent this will exclude the patients. This includes patients who unable to sit in a dark environment, have claustrophobic, inability to sit still for a few minutes
* Any other past medical, physiological or demographic concerns. This includes any patients with skin blemishes that are present at the dermis over the tumor, as these are of particular interest for use of this technique. This also includes open wounds on the area of interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants will be identified by a member of the patient's treatment team, the protocol investigator, or research team.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of clinical Cerenkov luminescence imaging by achieving satisfactory imaging at least a rate of 80% | Through study completion, an average of 24 hours
  The primary objective is to explore the overall feasibility of clinical Cerenkov imaging on patients with any tumors with nodal metastases (existing or suspected) scheduled for routine clinical FDG PET or 131I therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Grimm, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan - Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pratt EC, Skubal M, Mc Larney B, Causa-Andrieu P, Das S, Sawan P, Araji A, Riedl C, Vyas K, Tuch D, Grimm J. Prospective testing of clinical Cerenkov luminescence imaging against standard-of-care nuclear imaging for tumour location. Nat Biomed Eng. 2022 May;6(5):559-568. doi: 10.1038/s41551-022-00876-4. Epub 2022 Apr 11. PMID 35411113
- See also: Memorial Sloan Kettering Cancer Center — http://mskcc.org

DOCUMENTS (1):
  • Informed Consent Form (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/84/NCT03484884/ICF_000.pdf